CLINICAL TRIAL: NCT02387411
Title: High-intensity Interval Versus Combined High-intensity Interval and Strength Exercise Training in Chronic Heart Failure
Brief Title: High-intensity Interval Versus Combined Exercise Training in CHF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Athens (Other)
Responsible Party: Principal Investigator, Serafim Nanas, Prof Critical Care Medicine, University of Athens
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: not applied
Record Dates: First submitted 2015-02-19; First posted 2015-03-13 (Estimated); Last update posted 2015-03-13 (Estimated); Status verified 2015-03

CONDITIONS: Heart Failure
Keywords: heart failure; aerobic exercise; strength training; cardiopulmonary rehabilitation; high-intensity exercise training
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interval group (Active Comparator): high-intensity interval exercise training
  Interventions: Other: High-intensity interval exercise training
- Combined group (Active Comparator): combined exercise training
  Interventions: Other: Combined exercise training

INTERVENTIONS:
Other: High-intensity interval exercise training — High-intensity interval exercise training [4 reps * (4 min at 80% VO2peak + 3 min at 50% VO2peak)]
  Arms: Interval group
Other: Combined exercise training — High intensity [2 reps * (4 min at 80% VO2peak + 3 min at 50% VO2peak)] and strength exercise training (2-4 sets, 10-12 reps, 60-65% 1RM, for quadriceps and hamstrings, 14 min in total)
  Arms: Combined group

SUMMARY:
Chronic heart failure (CHF) is a clinical syndrome presented with central, cardiac deterioration as well as peripheral vascular and muscular abnormalities, resulting finally to reduced exercise tolerance, quality of life and mortality rates. Exercise training is a major component of rehabilitation / secondary prevention interventions, inducing significant beneficial changes in mechanisms of pathophysiology, exercise tolerance, functional capacity and quality of life, while a positive impact on hospitalization and mortality reduction should not be also excluded. There has been growing interest in the characteristics and modalities of exercise training able to induce optimal benefits. High intensity and interval mode have been shown to induce greater benefits than moderate intensity and continuous mode regimes. Additionally, there has been sound rationale for the inclusion of strength training, which has been also shown able to yield benefits in terms of exercise capacity and quality of life. However, there haven't been much data on the so called combined regimes, which include both aerobic exercise and strength training. This study aims at investigating the effects of combined high-intensity interval and strength training compared to high-intensity interval exercise alone in CHF.

ELIGIBILITY:
Inclusion Criteria:

* stable heart failure
* ejection fraction <=45%
* optimal medical treatment
* NYHA class <=III

Exclusion Criteria:

* contraindications for maximal cardiopulmonary exercise testing (CPET)
* moderate to severe COPD
* inability to follow exercise programs due to orthopaedic problems

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2010-05; Primary Completion 2015-06 (Estimated); Study Completion 2015-06 (Estimated)

PRIMARY OUTCOMES:
aerobic exercise capacity (assessed by cardiopulmonary exercise testing) | 3 months

SECONDARY OUTCOMES:
strength exercise capacity (assessed by 1-repetition maximum test) | 3 months
quality of life (assessed by MLWHF questionnaire) | 3 months
quadriceps local adaptations (assessed by muscle biopsies) | 3 months
quadriceps cross sectional area (assessed by CT) | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Serafim Nanas, MD, Prof., Study Chair — Cardiopulmonary Exercise Testing & Rehabilitation Laboratory, 1st Critical Care Dpt, School of Medicine, University of Athens, Greece
Locations (1):
- Cardiopulmonary Exercise Testing & Rehabilitation Laboratory, 1st Critical Care Dpt, School of Medicine, University of Athens, Athens, Greece

REFERENCES:
- [Derived] Tryfonos A, Tzanis G, Karatzanos Epsilon, Koutsilieris M, Nanas S, Philippou A. Inflammation- and Tissue Remodeling-Related Gene Responses in Skeletal Muscle of Heart Failure Patients Following High-Intensity Interval Training. Rev Cardiovasc Med. 2023 Feb 6;24(2):46. doi: 10.31083/j.rcm2402046. eCollection 2023 Feb. PMID 39077398
- [Derived] Alshamari M, Kourek C, Sanoudou D, Delis D, Dimopoulos S, Rovina N, Nanas S, Karatzanos E, Philippou A. Does the Addition of Strength Training to a High-Intensity Interval Training Program Benefit More the Patients with Chronic Heart Failure. Rev Cardiovasc Med. 2023 Jan 16;24(1):29. doi: 10.31083/j.rcm2401029. eCollection 2023 Jan. PMID 39076879
- [Derived] Tryfonos A, Tzanis G, Pitsolis T, Karatzanos E, Koutsilieris M, Nanas S, Philippou A. Exercise Training Enhances Angiogenesis-Related Gene Responses in Skeletal Muscle of Patients with Chronic Heart Failure. Cells. 2021 Jul 28;10(8):1915. doi: 10.3390/cells10081915. PMID 34440684